CLINICAL TRIAL: NCT00599651
Title: Randomized Controlled Trial of Surfactant Administration by Laryngeal Mask Airway (LMA)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was closed due to extremely low enrollment
Sponsor: University of Virginia (Other)
Collaborators: LMA North America (Unknown); ONY (Industry)
Responsible Party: John Kattwinkel, MD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11851
Record Dates: First submitted 2007-12-29; First posted 2008-01-24 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Respiratory Distress Syndrome; Newborn RDS
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome; Pulmonary Atelectasis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Surfactant by LMA
  Interventions: Device: Surfactant administered via Laryngeal Mask Airway (LMA)
- 2 (Other): Standard of care
  Interventions: Other: standard of care (nasal CPAP and supplemental oxygen)

INTERVENTIONS:
Device: Surfactant administered via Laryngeal Mask Airway (LMA) — Standard volume of Infasurf surfactant (3 mL/kg) will be injected in 2-4 aliquots into the proximal end of the LMA.
  Other Names: Infasurf; LMA
  Arms: 1
Other: standard of care (nasal CPAP and supplemental oxygen) — Standard of care will be utilized which may mean surfactant is administered
  Arms: 2

SUMMARY:
In this protocol we will conduct a randomized controlled trial where babies with respiratory distress syndrome (RDS) who have not yet reached criteria for intubation, will be randomized to receive surfactant by LMA or to continue receiving standard therapy of nasal CPAP and supplemental oxygen. All babies will be given surfactant by endotracheal tube if they reach "failure" criteria, which is the standard criterion for surfactant administration (i.e., FiO2= 65% while receiving nasal CPAP).

The objective of this RCT is to determine if surfactant can be successfully administered by LMA, thus perhaps avoiding the need for endotracheal intubation. The hypothesis is that fewer babies in the LMA group would reach failure criteria.

DETAILED DESCRIPTION:
Neonatal respiratory distress syndrome (RDS) is an illness of prematurity that results from insufficient surfactant in the lungs. Standard therapy for RDS is to place the baby in an oxygen hood or on nasal CPAP with supplemental oxygen, and if more than approximately 60% oxygen is required, an endotracheal tube is placed and a surfactant solution is injected into the tube.

An LMA is an FDA-approved, commercially-available device that is commonly used to substitute for an endotracheal tube.(1) The device consists of a tube, similar to an endotracheal tube, which has an inflatable donut-shaped cap at one end. The cap end of the LMA is placed through the mouth so that it lies over the larynx and the cap is then inflated. The opening of the tube is then proximal to the opening of the larynx and is sealed off from other structures that open into the pharynx (e.g., the esophagus). The other end of the LMA can then be attached to a resuscitation bag or mechanical ventilator to provide lung inflation.

This is a randomized controlled trial, where babies with moderate RDS, who have not received surfactant prophylaxis and have not yet required endotracheal intubation and who are large enough to accept an LMA, will be randomized either to receive surfactant by LMA or to be managed under standard protocol. Infants who weigh > 1200 gms and have been diagnosed with respiratory distress syndrome and have only minimal to moderate lung disease (i.e., currently receiving nasal CPAP and requiring 30-60% supplemental oxygen) will be eligible. After consent has been obtained, an envelope will be opened and the infant will be assigned to either the "LMA" or the "Standard" group.

Those in the "LMA" group will have an LMA inserted by routine technique, the cuff will be inflated, and the baby's respirations will be gently assisted with a flow-inflating anesthesia bag. When it is evident from physical examination and pulse oximetry that respiratory support is stable, the standard volume of Infasurf surfactant (3 mL/kg) will be injected in 2-4 aliquots into the proximal end of the LMA. Each aliquot will be followed by gentle positive-pressure assistance from the anesthesia bag until the surfactant has disappeared from the tube, and the infant will then be rotated to another position prior to the next aliquot. A minimum of both lateral positions will be used. After all aliquots have been administered, the LMA will be removed and the baby will be returned to nasal CPAP and managed by routine protocol. A baby in the LMA group may receive a subsequent LMA treatment if he/she requires a > 10 percentage-point increase in supplemental oxygen requirement for a > 30-minute period. Any subsequent dose cannot be given < 6 hours from a previous dose and a maximum of 3 total LMA doses may be given. No LMA surfactant may be administered under this protocol after 96 hours of age.

If a baby in either group reaches "failure" criteria, as described below, he/she will receive standard therapy for severe RDS, which involves endotracheal intubation and administration of surfactant by endotracheal tube. It is estimated that approximately half of the patients in the standard group will go on to reach the failure threshold.

"Failure" is defined as follows:

* FiO2 exceeding 65% for 15 minutes to achieve a consistent post-ductal oxygen saturation of 88-92%, OR
* Apnea of sufficient degree to warrant endotracheal intubation, OR
* Judgment by attending physician that endotracheal intubation is necessary. All subjects who reach failure criteria will receive endotracheal intubation and conventional surfactant therapy with Infasurf, unless considered contraindicated by the attending physician.

All patients will have FiO2 adjusted to maintain post-ductal oxygen saturation of 88-92% and will continue to receive nasal CPAP until either reaching failure criteria, or until FiO2 < 30%. If a subject does not reach failure criteria, nasal CPAP will be weaned to off and the baby will be place in an oxygen hood until FiO2 = room air. Babies may then be removed from the hood and returned to supplemental oxygen as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Birthweight > 1200 grams
* Chronologic age < 72 hours.
* Diagnosis of RDS by clinical and radiographic criteria.
* Treated with nasal CPAP and supplemental oxygen > 30% and not requiring > 60% FiO2 for longer than 30 minutes to maintain SaO2 88-95%.
* Parental consent.

Exclusion Criteria:

* Birthweight < 1200 gms.
* Diagnosis other than RDS (e.g., meconium aspiration syndrome).
* Babies who require or have already had endotracheal intubation.
* Babies with congenital anomalies or conditions thought by the attending physician to contribute to respiratory symptoms and/or to restrict adequate spontaneous breathing (e.g., congenital heart disease, obtundation from maternal drugs, certain airway malformations, diaphragmatic hernia).

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 380 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is reaching or not reaching failure criterion (FiO2= 65% while receiving nasal CPAP). | 96 Hours

SECONDARY OUTCOMES:
Duration of intubation | Birth to discharge
Nasal CPAP and requirement for supplemental oxygen | Birth to discharge
Time to reach full enteral feedings | Birth to discharge
Incidence of laryngeal edema | 96 hours
Duration of hospitalization | Birth to discharge

CONTACTS AND LOCATIONS:
Overall Officials: John Kattwinkel, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Abdel-Latif ME, Walker E, Osborn DA. Laryngeal mask airway surfactant administration for prevention of morbidity and mortality in preterm infants with or at risk of respiratory distress syndrome. Cochrane Database Syst Rev. 2024 Jan 25;1(1):CD008309. doi: 10.1002/14651858.CD008309.pub3. PMID 38270182